CLINICAL TRIAL: NCT00431808
Title: Randomized Controlled Trial to Evaluate the Safety and Immunogenicity of Recombinant Pichia Pastoris-Expressed P. Falciparum Apical Membrane Antigen 1 (PfAMA-1-FVO[25-545]) Versus Tetanus Toxoid, in Healthy Malian Adult in Bandiagara
Brief Title: Safety and Immunogenicity of Apical Membrane Antigen 1 (PfAMA-1-FVO[25-545])
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: African Malaria Network Trust (Network)
Responsible Party: Roma Chilengi, African Malaria Network Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AMA1_02_07; MU-08
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Malaria
Keywords: Malaria; vaccine; Apical Membrane Antigene; Mali; Adults
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I, AMA1 vaccine (Experimental): 20 volunteers will receive 3 doses of the vaccine
  Interventions: Biological: Malaria vaccine AMA1 (PfAMA-1-FVO[25-545]; Biological: AMA1

INTERVENTIONS:
Biological: Malaria vaccine AMA1 (PfAMA-1-FVO[25-545] — 3 doses of AMA 1 vaccine
Biological: AMA1 — 50 micrograms of AMA1

SUMMARY:
This study will be the first time that the candidate malaria vaccine Apical Membrane Antigen 1 (PfAMA-1-FVO[25-545]) will be tested in malaria endemic populations. The phase Ib study will include adults who will be randomly allocated to either receive the malaria vaccine or the vaccine against Tetanus. Each participant will receive 3 immunizations, without the clinical investigators or the participants themselves knowing what has been given. They will then be follow-up up for immediate reactions to vaccination, and also over a longer term of one year. Blood will be taken to evaluate the biological safety parameters and also immune responses.

DETAILED DESCRIPTION:
This will be a randomized controlled trial to evaluate the Safety and Immunogenicity of recombinant pichia pastoris blood stage malaria vaccine Apical Membrane Antigen 1 (PfAMA-1-FVO[25-545]) versus tetanus toxoid, in healthy Malian adults in Bandiagara.

A phase Ia trial is currently ongoing and its interim results will be used to select the best dose/adjuvant combination to be brought to Africa. The trial is evaluating safety and immunogenicity of AMA-1 (10 µg or 50 µg) adjuvanted with aluminum hydroxide or Montanide ISA 720, or ASO2.

* Primary objective:

  - To evaluate the safety of one dose of AMA-1 (10 µg or 50 µg) adjuvanted with aluminum hydroxide or Montanide ISA 720, or ASO2, given at D0, D28 and D56 in healthy Malian adults.
* Secondary Objectives:

  * To assess the humoral response to the vaccine antigen by measuring the variation in the level of IgG and its ability to recognize the native protein on merozoites.
  * To assess the cellular immune response by measuring the T cell proliferation and cytokine production following in vitro stimulation with the vaccine antigen.

The primary immunizations will be administered on days 0, 28 and a boost given at day 56. The participants will be followed up actively during the vaccination phase, and passively for one another 9 months. The will be 19 scheduled clinic visits and following will the the schedule for obtaining serology data D-28, D0, D28, D56, D84, D140 and D365

* The primary evaluation will include the following:

  * Solicited adverse events measured from day 0 to day 7 after each dose;
  * Unsolicited adverse events measured up to one month after each dose;
  * Serious Adverse Event (SAE) measured during the 12 months of study duration.
  * Biological safety: two and four weeks after each vaccination, and thereafter every 12 weeks, in reference with the baseline before the first dose, by measuring the following RBC, hemoglobin, hematocrit, MCV, MCH, MCHC, platelets, WBC with differential counts, potassium, sodium, ASAT, ALAT, total bilirubin, alkaline phosphatase, γGT, creatinin.
* Secondary evaluation criteria:

  * The humoral response to the vaccine antigen: assessed by measuring the level of IgG by ELISA.
  * An IFA for at least two parasite strains will be used to verify that the antibodies elicited by the vaccine recognize the native protein on merozoites
* Statistical methods:

Descriptive methods shall be employed to evaluate the above criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years inclusive at the time of screening
* Residing in Bandiagara for the duration of the study
* Separate written informed consent obtained before screening and study start, respectively
* Available to participate in follow-up for the duration of study (14 months)
* General good health based on history and clinical examination
* Willingness not to become pregnant during the first five months of the study for female participants

Exclusion Criteria:

* Previous vaccination with a investigational vaccine or a rabies vaccine
* Use of a investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first study immunization, or planned use up to 30 days after the third immunization
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first immunization. This includes any dose level of oral steroids or inhaled steroids, but not topical steroids
* Confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* Confirmed or suspected autoimmune disease
* History of allergic reactions or anaphylaxis to immunizations or to any vaccine component
* History of serious allergic reactions to any substance, requiring hospitalization or emergent medical care
* History of allergy to vaccines components
* History of splenectomy
* Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25 times the upper limit of normal of the testing laboratory).
* Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory, or more than trace protein or blood on urine dipstick testing).
* Laboratory evidence of hematologic disease (absolute leukocyte count <4000/mm3 or >14,500/mm3, absolute lymphocyte count <1500/mm3, platelet count <120,000/mm3, or hemoglobin <10.0 g/dL).
* Administration of immunoglobulins and/or any blood products within the three months preceding the first study immunization or planned administration during the study period.
* Simultaneous participation in any other interventional clinical trial
* Acute or chronic pulmonary, cardiovascular, hepatic, renal or neurological condition, malnutrition, or any other clinical findings that in the opinion of the PI may increase the risk of participating in the study
* Other condition that in the opinion of the PI would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
*Safety evaluation through: | 1 year
Solicited adverse events measured from day 0 to day 7 after each dose; | 7 days
Unsolicited adverse events measured up to one month after each dose; | 84 days
Serious Adverse Events measured during the 12 months of study duration. | 1 year
Biological safety: two and four weeks after each vaccination, and thereafter every 12 weeks, in reference with the baseline before the first dose, by measuring the following : | 1 year
RBC, hemoglobin, hematocrit, MCV, MCH, MCHC, platelets, WBC with differential counts, potassium, sodium, ASAT, ALAT, total bilirubin, alkaline phosphatase, γGT, creatinin | 1 year

SECONDARY OUTCOMES:
*Immunogenicity evaluation through: | 84 days
The humoral response to the vaccine antigen: assessed by measuring the level of IgG by ELISA. | 84 days
An IFA for at least two parasite strains will be used to verify that the antibodies elicited by the vaccine recognize the native protein on merozoites. | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Mahamadou A Thera, MD MPH, Principal Investigator — Malaria Research and Training Center
Locations (1):
- Malaria Research and Training Center, Bandiagara, Mali

REFERENCES:
- [Derived] Thera MA, Coulibaly D, Kone AK, Guindo AB, Traore K, Sall AH, Diarra I, Daou M, Traore IM, Tolo Y, Sissoko M, Niangaly A, Arama C, Baby M, Kouriba B, Sissoko MS, Sagara I, Toure OB, Dolo A, Diallo DA, Remarque E, Chilengi R, Noor R, Sesay S, Thomas A, Kocken CH, Faber BW, Imoukhuede EB, Leroy O, Doumbo OK. Phase 1 randomized controlled trial to evaluate the safety and immunogenicity of recombinant Pichia pastoris-expressed Plasmodium falciparum apical membrane antigen 1 (PfAMA1-FVO [25-545]) in healthy Malian adults in Bandiagara. Malar J. 2016 Aug 30;15(1):442. doi: 10.1186/s12936-016-1466-4. PMID 27577237